CLINICAL TRIAL: NCT06548971
Title: Safety and Efficacy of Treatment With Early Antiplatelet Administration After Intravenous Thrombolysis for Acute Ischemic Stroke (TREND-IVT): A Multicenter, Randomized, Placebo-controlled, Clinical Trial
Brief Title: Early Antiplatelet Administration After Intravenous Thrombolysis for Acute Ischemic Stroke (TREND-IVT)
Acronym: TREND-IVT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TREND-IVT
Record Dates: First submitted 2024-08-03; First posted 2024-08-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke; Cerebral Infarction
Keywords: Acute ischemic stroke; Intravenous thrombolysis; Early neurological deterioration; Aspirin
MeSH Terms: conditions — Ischemic Stroke; Cerebral Infarction | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Patients in the interventional group will receive early antiplatelet treatment with oral aspirin within 3 hours of initiating intravenous thrombolysis. In addition, the best medical management will be administered according to the guidelines.
  Interventions: Drug: Aspirin; Other: Best medical management
- Control group (Placebo Comparator): Patients in the control group will receive placebos within 3 hours of initiating intravenous thrombolysis. In addition, the best medical management will be administered according to the guidelines.
  Interventions: Drug: Placebo; Other: Best medical management

INTERVENTIONS:
Drug: Aspirin — Patients in the interventional group will chew 300mg of aspirin enteric-coated tablets as soon as possible after randomization. If swallowing difficulties arise, the tablets can be crushed and administered via a nasogastric tube.
  Arms: Interventional group
Drug: Placebo — Patients in the control group will chew 300mg of placebos as soon as possible after randomization. If swallowing difficulties arise, the placebo can be crushed and administered via a nasogastric tube.
  Arms: Control group
Other: Best medical management — Patients in both groups will receive the best medical management according to the guidelines.

SUMMARY:
Stroke is the second leading cause of death worldwide, and ischemic stroke is the most frequent type. Intravenous thrombolysis with recombinant tissue plasminogen activator within 4.5 hours of symptom onset is the most effective therapy for patients with acute ischemic stroke. However, ischemic stroke progression and early reocclusion are not an uncommon phenomenon in patients after intravenous thrombolysis, resulting in neurological deterioration, which is associated with unfavorable functional outcomes. The underlying mechanism mainly involves the augmented platelet activation, triggered by the activated coagulation cascade during thrombolysis, which peaks within 2 hours of initiating rt-PA administration. Therefore, early antiplatelet therapy following intravenous thrombolysis represents a promising therapeutic approach to prevent neurological deterioration and improve the functional outcome of patients treated with intravenous thrombolysis.

Currently, guidelines recommend initiating antiplatelet therapy 24 hours after intravenous thrombolysis due to the potential risk of increased bleeding. The safety and efficacy of early antiplatelet treatment following intravenous thrombolysis in patients with acute ischemic stroke remain clear.

The study aims to test the hypothesis that in patients with acute ischemic stroke treated with intravenous thrombolysis, early administration of oral aspirin will improve functional outcomes without increasing the risk of intracranial hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Acute ischemic stroke treated with intravenous thrombolysis with alteplase or tenecteplase within 4.5 hours of onset or time last known well, and can receive the study drug treatment within 3 hours of initiating intravenous thrombolysis.
3. Residual NIHSS score > 5 points assessed 1 hour after initiation of intravenous thrombolysis and prior to randomization.
4. Informed consent obtained from patients or an authorized representative.

Exclusion Criteria:

1. Stroke caused by definite large vessel occlusion (including A1/A2 segments of the anterior cerebral artery, M1/M2 segments of the middle cerebral artery, P1/P2 segments of the posterior cerebral artery, intracranial/extracranial segments of the internal carotid artery, basilar artery, and bilateral vertebral artery occlusion) confirmed by vessel imaging (including computed tomography angiography [CTA] or magnetic resonance angiography [MRA]), or scheduled for endovascular treatment (including mechanical thrombectomy, intra-arterial thrombolysis, and angioplasty).
2. Intracranial hemorrhage confirmed by imaging post-thrombolysis.
3. Definite or suspected cardioembolic stroke.
4. Stroke caused by other determined causes, including nonatherosclerotic vasculopathies (moyamoya disease, artery dissection, arteritis), hypercoagulable states, or hematological disorders.
5. Use of antiplatelet therapy within one week prior to stroke onset, novel anticoagulant drugs within 48 hours prior to stroke onset, or treatment with warfarin with an international normalized ratio (INR)>1.7.
6. Prior history of moderate or severe ischemic stroke events with residual neurological disability.
7. Pre-stroke mRS score > 1.
8. Severe consciousness disturbance with NIHSS item 1a (level of consciousness) ≥ 2 points.
9. Post-thrombolysis imaging indicates an infarct area larger than 1/2 responsible artery supply area.
10. Known contraindications for antiplatelet therapy, such as coagulation disorders, or systemic bleeding
11. History of aspirin allergy.
12. Anticipated indications for anticoagulant therapy during the study period (e.g., atrial fibrillation, mechanical heart valve, deep vein thrombosis, pulmonary embolism, antiphospholipid syndrome, hypercoagulable state)
13. Presence of malignant tumors, chronic hemodialysis, severe renal insufficiency (GFR < 30 mL/min or serum creatinine > 220 μmol/L [2.5 mg/dL]), severe hepatic insufficiency (serum alanine aminotransferase [ALT] >2 times the upper limit of normal, or serum aspartate aminotransferase [AST] >2 times the upper limit of normal), severe heart failure (New York Heart Association [NYHA] Functional Classification Class III or IV)
14. Severe non-cardiovascular complications with an expected survival of less than 6 months.
15. Unavailability for follow-up.
16. Presence of dementia, psychiatric disorders, or other known neurological conditions that complicate follow-up.
17. Current participation in another therapeutic study with ongoing treatment and follow-up.
18. Other conditions that make the patient unsuitable for participation in the study as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1184 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a modified Rankin scale (mRS) score of 0-1 at 90-day follow up. | Ninety days after stroke.
  The mRS ranges from 0 to 6, with higher scores indicating a worse outcome. The primary outcome measure is based on the mRS score, which is dichotomized to define the excellent functional outcome as mRS score of 0-1 at 90-days follow up.

SECONDARY OUTCOMES:
The proportion of patients with a modified Rankin scale (mRS) score of 0-1 at 30-day follow up. | Thirty days after stroke.
  The mRS ranges from 0 to 6, with higher scores indicating a worse outcome. The primary outcome measure is based on the mRS score, which is dichotomized to define the excellent functional outcome as mRS score of 0-1 at 30-days follow up.
The proportion of patients with a modified Rankin scale (mRS) score of 0-2 at 90-day follow up. | Ninety days after stroke.
  The mRS ranges from 0 to 6, with higher scores indicating a worse outcome. Functional independence is defined as mRS of 0-2.
The shift analysis in the 90-day modified Rankin scale (mRS) score. | Ninety days after stroke.
  The mRS ranges from 0 to 6, with higher scores indicating a worse outcome.
The proportion of patients achieving neurological improvement. | Within 48 hours after stroke.
  Neurological improvement is defined as a decrease of ≥2 points in the NIHSS score at 48 hours of randomization compared to baseline assessment.
The proportion of patients experiencing early neurological deterioration. | Within 24 hours after stroke.
  Early neurological deterioration is defined as an increase of ≥4 points in the NIHSS score within 24 hours of randomization compared with the minimum NIHSS score before deterioration.
The changes in the NIHSS score at 24 hours, 48 hours, and 7 days of enrollment as compared with the baseline. | Within 7 days after stroke.
  The NIHSS ranges from 0 to 42 points, with higher scores indicating worse neurological deficits.

OTHER OUTCOMES:
Incidence of symptomatic intracranial hemorrhage. | Within 48 hours after stroke.
  Symptomatic intracranial hemorrhage is defined as the demonstration of hemorrhage within brain parenchyma on head imaging leading to an increase of at least 4 points in the NIHSS score, according to the criteria of the European Cooperative Acute Stroke Study III (ECASS III).
Incidence of any intracranial hemorrhage. | Within 48 hours after stroke.
  Any intracranial hemorrhage is defined as the demonstration of hemorrhage within brain parenchyma on head imaging, according to the criteria of the ECASS III.
Incidence of systemic hemorrhage. | Within 90 days after stroke.
  The incidence of systemic hemorrhage at any time from randomization through day 90, according to the criteria of the GUSTO.
Incidence of recurrent stroke or other vascular events. | Within 90 days after stroke.
  The incidence of recurrent stroke or other vascular events (including hemorrhagic and ischemic stroke, myocardial infarction, and cardiovascular death) within 90 days of randomization.
All-cause death. | Within 90 days after stroke.
  The incidence of death events at any time from randomization through day 90.
Incidence of Adverse Events/Serious Adverse Events | Within 90 days after stroke.
  The incidence of other adverse events and serious adverse events at any time from randomization through day 90.

CONTACTS AND LOCATIONS:
Locations (71):
- China (71):
  - The Third The People's Hospital Of Bengbu, Bengbu, Anhui
  - Suzhou municipal hospital, Suzhou, Anhui
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Aerospace central hospital, Haidian, Beijing Municipality
  - Beijing Pinggu District Hospital, Pinggu, Beijing Municipality
  - Beijing Luhe Hospital affiliated to Capital Medical University, Tongzhou, Beijing Municipality
  - Fujian university affiliated provincial hospital, Fuzhou, Fujian
  - The First Affiliated Hospital Of Xiamen University, Xiamen, Fujian
  - Xiamen Xinglin hospital, Xiamen, Fujian
  - Zhangzhou Hospital of Fujian Province, Zhangzhou, Fujian
  - Brain Hospital Affiliated to Guangzhou Medical University, Guangzhou, Guangdong
  - Guigang people's hospitalv, Guigang, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi
  - The Second Affiliated Hospital of Guizhou Medical University, Kaili, Guizhou
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Cangzhou combination of Chinese traditional and western medicine hospital, Cangzhou, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hejian city People's Hospital, Cangzhou, Hebei
  - Handan Central Hospital, Handan, Hebei
  - Handan first hospital, Handan, Hebei
  - The First Hospital Of Qiqihar, Qiqihar, Heilongjiang
  - Hua county People's Hospital, Anyang, Henan
  - Jun county people's hospital, Hebi, Henan
  - Jiaozuo Second People's Hospital, Jiangzuo, Henan
  - First People's Hospital of Luoyang, Luoyang, Henan
  - Luoyang Yanshi People's Hospital, Luoyang, Henan
  - Nanyang nanshi hospital, Nanyang, Henan
  - Huanghe Sanmenxia hospital, Sanmenxia, Henan
  - Shangqiu Third People's Hospital, Shangqiu, Henan
  - Shangqiu First People's Hospital, Shangqiu, Henan
  - Ningling county people's hospital, Shangqucun, Henan
  - Xihua People's Hospital, Zhoukou, Henan
  - Luyi county people's hospital, Zhoukou, Henan
  - Zhumadian Central Hospital, Zhumadian, Henan
  - The Third People's Hospital of Hubei Province, Hainan, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - Changde Taoyuan County People's Hospital, Changde, Hunan
  - Chenzhou first people's hospital, Chenzhou, Hunan
  - Liuyang Jili Hospital, Guankou, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Affiliated Hospital of Inner Mongolia University for the Nationalities, Tongliao, Inner Mongolia
  - Ulanqab Central Hospital, Ulanqab, Inner Mongolia
  - Zha Lan Tun Shi Zhong Meng Yi Yuan, Zhalantun, Inner Mongolia
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Fourth Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jingdezhen NO.1 People's Hospital, Jingdezhen, Jiangxi
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Anshan Changda hospital, Anshan, Liaoning
  - Donggang city Central Hospital, Dandong, Liaoning
  - Fushun Mining Bureau General Hospital, Fushun, Liaoning
  - Togtoh county hospital, Neimeng, Neimeng
  - Dongying people's hospital, Dongying, Shandong
  - Shengli oilfield central hospital, Dongying, Shandong
  - Shandong province qianfoshan hospital, Jinan, Shandong
  - Jinan Third People's Hospital, Jinan, Shandong
  - Liaocheng people's hospital, Liaocheng, Shandong
  - The Third People Hospital In Liaocheng, Liaocheng, Shandong
  - Gaotang county people's hospital, Liaocheng, Shandong
  - Pingdu city traditional Chinese medicine hospital, Qingdao, Shandong
  - Juxian county people's hospital, Rizhao, Shandong
  - Rizhao traditional Chinese medicine hospital, Rizhao, Shandong
  - Shandong health group feicheng hospital, Taian, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Weinan central hospital, Weinan, Shanxi
  - Shenzhen Second People's Hospital, Shenzhen, Shenzhen
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Ya 'an People's Hospital, Ya'an, Sichuan
  - Shihezi City People's Hospital, Shihezi, Xinjiang
  - Haiyan People's Hospital, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] Demaerschalk BM, Kleindorfer DO, Adeoye OM, Demchuk AM, Fugate JE, Grotta JC, Khalessi AA, Levy EI, Palesch YY, Prabhakaran S, Saposnik G, Saver JL, Smith EE; American Heart Association Stroke Council and Council on Epidemiology and Prevention. Scientific Rationale for the Inclusion and Exclusion Criteria for Intravenous Alteplase in Acute Ischemic Stroke: A Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Feb;47(2):581-641. doi: 10.1161/STR.0000000000000086. Epub 2015 Dec 22. PMID 26696642
- [Background] Wu C, Sun C, Wang L, Lian Y, Xie N, Huang S, Zhao W, Ren M, Wu D, Ding J, Song H, Wang Y, Ma Q, Ji X. Low-Dose Tirofiban Treatment Improves Neurological Deterioration Outcome After Intravenous Thrombolysis. Stroke. 2019 Dec;50(12):3481-3487. doi: 10.1161/STROKEAHA.119.026240. Epub 2019 Oct 1. PMID 31570084
- [Background] Zinkstok SM, Roos YB; ARTIS investigators. Early administration of aspirin in patients treated with alteplase for acute ischaemic stroke: a randomised controlled trial. Lancet. 2012 Aug 25;380(9843):731-7. doi: 10.1016/S0140-6736(12)60949-0. Epub 2012 Jun 28. PMID 22748820
- [Background] Zhao W, Li S, Li C, Wu C, Wang J, Xing L, Wan Y, Qin J, Xu Y, Wang R, Wen C, Wang A, Liu L, Wang J, Song H, Feng W, Ma Q, Ji X; TREND Investigators. Effects of Tirofiban on Neurological Deterioration in Patients With Acute Ischemic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2024 Jun 1;81(6):594-602. doi: 10.1001/jamaneurol.2024.0868. PMID 38648030